CLINICAL TRIAL: NCT06082518
Title: Improving Post COVID-19 Syndrome With Hyperbaric Oxygen Treatments (PCS-HBOT Study)
Brief Title: Improving Post COVID-19 Syndrome With Hyperbaric Oxygen Treatments
Acronym: PCS-HBOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5825
Record Dates: First submitted 2023-09-11; First posted 2023-10-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Post COVID-19 Condition; Post-COVID-19 Syndrome; Post-COVID Syndrome; COVID-19; Fatigue; Fatigue Syndrome, Chronic
Keywords: Hyperbaric Oxygen Therapy; HBOT; Post COVID-19 Condition; Fatigue; Severe Acute Respiratory Syndrome-CoV-2; COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Fatigue; Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Specialist hyperbaric physicians, blinded to group allocation, will provide treatment and follow patients daily throughout their treatment course.
  Outcomes Assessor will also be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immediate start of hyperbaric treatments (Experimental): HBOT treatments will be scheduled to start immediately after referral.
  Interventions: Device: Monoplace Hyperbaric Chamber (Class III medical device).
- Delayed start of hyperbaric treatments (Experimental): HBOT treatments will be scheduled to start 60 days after referral.
  Interventions: Device: Monoplace Hyperbaric Chamber (Class III medical device).

INTERVENTIONS:
Device: Monoplace Hyperbaric Chamber (Class III medical device). — 40 hyperbaric oxygen therapy (HBOT) treatments (90 minute exposures at 2 atmospheres (ATM) per treatment), scheduled daily from Monday to Friday (i.e., 5 treatments per week) until treatments are completed (approximately 8 weeks). Treatments will be delivered in a medical grade, Health Canada-approved monoplace hyperbaric chamber and overseen by specialist hyperbaric physicians and a Certified Hyperbaric Technologist.
  Device is being used in manner consistent with approved usage in Canada.

SUMMARY:
Over 500 million people have been infected with COVID-19, and to date, more than 6 million people have died. Many individuals who have recovered from COVID-19 continue to experience symptoms even after they have been "cured" of the disease. This condition is known as post COVID-19 condition, which can have serious health consequences. A common symptom among these individuals is chronic fatigue, characterized by persistent tiredness or lack of energy. This study aims to explore a novel treatment for symptoms of post COVID-19 condition, known as hyperbaric oxygen therapy. This approach has shown promise in helping people with post COVID-19 conditions and treating some other causes of fatigue.

Hyperbaric oxygen therapy involves placing patients in a small chamber where they receive high oxygen gas levels. However, this treatment is expensive and time-consuming, and it is unclear if this treatment can be effectively assessed in a large-scale research study. This small study will help us decide if conducting a large research study is feasible. The investigators aim to assess if hyperbaric oxygen therapy can improve symptoms of post COVID-19 condition, such as fatigue.

DETAILED DESCRIPTION:
Over 500 million individuals worldwide have contracted COVID-19. Among those that have 'recovered' from the acute infection, many suffer from post-COVID-19 condition (experiencing 1 or more symptoms 3 months from the onset of acute COVID-19 infection, with symptoms lasting at least 2 months). Many of these common symptoms, including fatigue, myalgia, and difficulty focusing ('brain fog'), can seriously compromise one's quality of life.

Existing treatments predominantly focus on supportive management and specific symptom control, and most approaches have mixed or limited effectiveness. Recently, hyperbaric oxygen therapy (HBOT), acknowledged for its anti-inflammatory effects, has emerged as a potential treatment for post-COVID-19 condition symptoms. However, HBOT is time and resource-intensive, requiring between 20-40 daily treatments. Therefore, the feasibility of assessing HBOT efficacy via a large-scale randomized controlled trial is still being determined. Hence, this study aims to evaluate adherence to the protocol and the feasibility of proceeding with the full trial. The goal of the full trial will be to evaluate the impact of HBOT treatment on post-COVID-19 condition symptoms.

This prospective, crossover, randomized pilot trial enrolls adult patients officially diagnosed with post-COVID-19 condition by a healthcare practitioner who continue to experience symptoms, particularly fatigue, at least 3 months following their initial COVID-19 infection. Participants will be assigned randomly (stratified by sex) to either begin HBOT treatments immediately or after a 60-day interval. All patients will be followed for 12 months from the start of treatment, with assessments at the time of enrollment (baseline), start of treatment (if starting 60 days after enrollment), 4 weeks after the start of treatment, and every 2 months from the first HBOT treatment for 1 year. A subjective questionnaire regarding patient satisfaction will also be completed after the last HBOT treatment session and at 1 year after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Officially diagnosed with post COVID-19 condition by a healthcare practitioner
3. At least three months since SARS-CoV-2 infection
4. Symptoms that persist more than 12 weeks:

   * Chronic fatigue (must include) along with one of the following symptoms:
   * Difficulty thinking or problem solving ('brain fog')
   * Stress or anxiety

Exclusion Criteria:

1. Contraindications/medically unfit to receive hyperbaric treatments at an outpatient facility (pneumothorax, in-patients, requiring infusions to maintain hemodynamics, active and unstable coronary disease)
2. Patients with cognitive difficulties and/or mental retardation before COVID diagnosis
3. History of traumatic brain injury
4. Unlikely to comply with follow-up assessments (e.g. no fixed address, plans to move out of town)
5. Known pregnancy or planning a pregnancy in women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate - referral | 9 months
  Quantify referral rate from healthcare providers
Recruitment rate - inclusion | 9 months
  Number of patients meeting inclusion criteria
Recruitment rate - consent | 9 months
  Patient consent rate
Adherence to HBOT protocol | 9 months recruitment + 8 weeks treatment
  Number of Participants received minimum 4 treatments per week with >35 treatments
Adherence to HBOT protocol - satisfaction | After last HBOT treatment and at 12 month follow-up
  Subjective patient satisfaction questionnaire inquiring about HBOT experience, barriers to and promoters of treatment
Feasibility of Clinical Outcome Measures | Up to 1 year after start of treatment
  Feasibility of implementation of clinical outcome scales (PDQ, FSS, SF-36) to be completed at the time of enrollment (baseline), start of treatment (if starting 60 days after enrollment), 4 weeks after the start of treatment, and every 2 months from the first HBOT treatment for 1 year.

SECONDARY OUTCOMES:
The impact of HBOT on post COVID-19 condition - PDQ | Up to 1 year after start of treatment
  The validated clinical deficit scale, Perceived Deficits Questionnaire (PDQ), will be used at the time of enrollment (baseline), start of treatment (if starting 60 days after enrollment), 4 weeks after the start of treatment, and every 2 months from the first HBOT treatment for 1 year
The impact of HBOT on post COVID-19 condition - FSS | Up to 1 year after start of treatment
  The validated clinical deficit scale, Fatigue Severity Scale (FSS), will be used at the time of enrollment (baseline), start of treatment (if starting 60 days after enrollment), 4 weeks after the start of treatment, and every 2 months from the first HBOT treatment for 1 year
The impact of HBOT on post COVID-19 condition - SF-36 | Up to 1 year after start of treatment
  The validated clinical deficit scale, QoL Short Form Survey (SF-36), will be used at the time of enrollment (baseline), start of treatment (if starting 60 days after enrollment), 4 weeks after the start of treatment, and every 2 months from the first HBOT treatment for 1 year.
The impact of time to initiation of HBOT on outcomes following initial infection outcome - PDQ | Up to 1 year after start of treatment
  Validated clinical deficit scales PDQ will be compared with FSS and SF-36 between immediate and delayed start groups
The impact of time to initiation of HBOT on outcomes following initial infection outcome - FSS | Up to 1 year after start of treatment
  Validated clinical deficit scale FSS will be compared with PDQ and SF-36 between immediate and delayed start groups
The impact of time to initiation of HBOT on outcomes following initial infection outcome - SF-36 | Up to 1 year after start of treatment
  Validated clinical deficit scale SF-36 will be compared with PDQ and FSS between immediate and delayed start groups
Initial infection severity as a mediator of HBOT impact - PDQ | Up to 1 year after start of treatment
  Validated clinical deficit scale PDQ will be compared relative to baseline scores
Initial infection severity as a mediator of HBOT impact - FSS | Up to 1 year after start of treatment
  Validated clinical deficit scale FSS will be compared relative to baseline scores
Initial infection severity as a mediator of HBOT impact - SF-36 | Up to 1 year after start of treatment
  Validated clinical deficit scale SF-36 will be compared relative to baseline scores
Long-term symptomatic impact at 1 year - PDQ | 12 month follow-up
  Assessed using validated clinical deficit scale PDQ at 12 months after start of treatment
Long-term symptomatic impact at 1 year - FSS | 12 month follow-up
  Assessed using validated clinical deficit scale FSS at 12 months after start of treatment
Long-term symptomatic impact at 1 year - SF-36 | 12 month follow-up
  Assessed using validated clinical deficit scales SF-36 at 12 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alam, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Jordan Tarshis, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request to study PIs following publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication, no limit on time.
Access Criteria: Contact directly study principal investigators.